CLINICAL TRIAL: NCT04531202
Title: Clinical Characterization Protocol for Severe Emerging Infections: Coronavirus
Brief Title: CORE Study COVID-19
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: D'Or Institute for Research and Education (Other)
Responsible Party: Sponsor
Other Study IDs: 29496920.8.0000.5262
Record Dates: First submitted 2020-08-26; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Coronavirus Infection (COVID-19)
Keywords: coronavirus
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with confirmed or suspected of coronavirus infe: Clinical and laboratory data will be collected throughout the acute illness period. Research data will be integrated with information available from hospital and regulatory files.

SUMMARY:
This is a Brazilian version of the Clinical Characterization Protocol for Serious Emerging Infections (ISARIC/WHO ). This is a standardized protocol for the rapid, coordinated clinical investigation of Coronavirus disease (COVID-19). Patients with acute illness suspected to be caused by emerging will be enrolled. This protocol has been designed to enable data to be prospectively collected.

DETAILED DESCRIPTION:
The study will be conducted at multiple sites (to be determined by the spread of disease and availability of resources). It is appreciated that settings will vary in terms of clinical infrastructure, resources and capacity. This study will enrol eligible patients (adults) with confirmed or suspected infection with a pathogen relevant to the study objectives. Recruitment of patients with Day 1 (enrolment) data and biological samples is the priority.

Observational analyses will be stratified according to available data. Outcome data for primary and secondary objectives will be derived from data from routine clinical and laboratory assessments performed as part of standard inpatient medical management at the treating site, documented using proportionate case report forms (CRF; either paper or web-based electronic 'eCRF'). Clinical and laboratory data will be collected throughout the acute illness period according to local resources. Priority at all times will be given to the collection of clinical information. Research data will be integrated as much as possible with information available from hospital and regulatory files.

ELIGIBILITY:
Inclusion Criteria:

* Suspected or proven Coronavirus infection (COVID-19)

Exclusion Criteria:

* Confirmed diagnosis of a pathogen unrelated to the objectives of this study (or other non-infectious diagnosis) and no indication or likelihood of co-infection with a relevant pathogen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with coronavirus infection and molecular laboratory diagnosis of COVID-19, made from material collected from the upper respiratory tract (nasopharynx or oropharynx) or from the lower respiratory tract (sputum, tracheal aspirate or bronchoalveolar lavage)
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-03-02 (Actual); Primary Completion 2020-09-30 (Estimated); Study Completion 2021-09-30 (Estimated)

PRIMARY OUTCOMES:
Clinical characterization of coronavirus disease-2019 (COVID-19) | 1 year
  Describe the clinical features of the illness or syndrome and complications, and determinants of severity.
  Assessment daily for 14 days, then hospital discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Bozza, phD, Principal Investigator — D'Or Institute for Research and Education (IDOR)
Locations (1):
- D'Or Institute for Research and Education (IDOR), Rio de Janeiro, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Dunning JW, Merson L, Rohde GGU, Gao Z, Semple MG, Tran D, Gordon A, Olliaro PL, Khoo SH, Bruzzone R, Horby P, Cobb JP, Longuere KS, Kellam P, Nichol A, Brett S, Everett D, Walsh TS, Hien TT, Yu H, Zambon M, Ruiz-Palacios G, Lang T, Akhvlediani T; ISARIC Working Group 3, ISARIC Council; Hayden FG, Marshall J, Webb S, Angus DC, Shindo N, van der Werf S, Openshaw PJM, Farrar J, Carson G, Baillie JK. Open source clinical science for emerging infections. Lancet Infect Dis. 2014 Jan;14(1):8-9. doi: 10.1016/S1473-3099(13)70327-X. No abstract available. PMID 24355025